CLINICAL TRIAL: NCT06298201
Title: Investigating of Effects of e-Based Physical Exercise in Patients With Multiple Sclerosis and Comorbidity
Brief Title: E-Based Physical Exercise in Patients With Multiple Sclerosis and Comorbidity
Acronym: COMPACT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IMAGINE2024
Record Dates: First submitted 2024-02-20; First posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-02

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; Comorbidity; physical exercise; e-Based
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial (RCT) with prospective longitudinal follow up
Who Masked: Participant
Masking Description: Due to the nature of the intervention, it is not feasible to blind participants or physiotherapists delivering the program. Nonetheless, to preserve the integrity of the trial, outcome assessors (researchers) will remain blinded to the allocation of treatments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E-Based Physical Exercise Intervention (Experimental): A randomized controlled trial (RCT) aimed at evaluating the effects of an e-based PE intervention at home in addition to conventional PE on the disability progression of pwMS comorbid conditions.
  Interventions: Other: E-Based Physical Exercise Intervention
- Conventional Physical Exercise (No Intervention): Conventional Physical Exercise will receive no e-based PE intervention

INTERVENTIONS:
Other: E-Based Physical Exercise Intervention — The intervention comprises a 6-months home-based resistance training for the lower extremities, conducted twice weekly.
  Arms: E-Based Physical Exercise Intervention

SUMMARY:
Background: Physical exercise (PE) improves symptoms and quality of life in patients with multiple sclerosis (pwMS). Comorbidity is prevalent among pwMS and may contribute to disease progression. Integrating and sustaining PE is challenging and E-based PE solutions have been proposed as a tool to support the integration of PE into daily life.

Aims: To assess the effect of e-based PE in addition to usual care in pwMS on clinical outcome and the levels of inflammatory, metabolic, and neurodegenerative mediators. Furthermore, to determine whether PE plays a role in the modification of comorbidities with a focus on vascular comorbidity and related risk factors, i.e., type 2 diabetes mellitus.

Method: This study will be prospective with longitudinal follow-up of pwMS with and without comorbidities. The physical activity of pwMS will be measured at baseline and after six months by accelerometers. In a randomized controlled trial (RCT) patients will be randomly assigned in a 1:1 ratio to receive either usual care or usual care plus an e-based PE program. The exercise program consists of resistance training with resistance bands targeting the lower extremities, including leg press, knee extension, hip flexion, hamstring curl, and hip extension. The sessions will enable participants to engage in group exercises from their homes through a secure online platform, supervised virtually by physiotherapists. The primary endpoints are walking capacity using the 6-meter walk test and the NEDA-3 scale, focusing on the absence of clinical relapses and disease progression, as indicated by an increase in the Expanded Disability Status Scale score and the absence of new disease activity on MRI (including new T2 lesions or enhancing lesions). Secondary outcomes will encompass measures of quality of life and fatigue, as well as levels of potential biomarkers like neurofilament light chain in blood and cerebrospinal fluid.

Conclusion: This study will contribute to the rehabilitation and improved quality of life of pwMS particularly of patients with comorbidities. The potential for e-based PE at home to encourage sustained exercise engagement among pwMS will be evaluated, offering a significant contribution to the field of digital healthcare solutions.

DETAILED DESCRIPTION:
Background Multiple sclerosis (MS) is an inflammatory demyelinating disease of the central nervous system (CNS). MS is a potentially disabling disease and occurs as a consequence of immune attacks on myelin and nerve fibers and may lead to neuronal damage (neurodegeneration) and consequently to the clinical accumulation of neurological disability. Over the last two decades, the age-specific prevalence of people with MS (pwMS) has increased, and aging may amplify the risk of comorbidities and conversion to a progressive disease course. Emerging evidence underscores the high prevalence of comorbidity in pwMS, evident even at the time of MS diagnosis. Comorbidities can lead to delayed MS diagnosis, accelerated disease progression, and diminished efficacy and safety of MS treatments, subsequently increasing mortality. Vascular comorbidities, in particular, are prevalent among MS patients, with risk factors including type 2 diabetes mellitus (T2DM), obesity, hyperlipidemia and hypertension.

Physical exercise (PE) is advocated as an effective treatment for at least 26 chronic diseases, including MS. In pwMS, PE has been shown to positively modulate peripheral inflammatory markers such as Tumour Necrosis Factor alpha (TNF alpha), interferon-gamma, Interleukin-4, interleukin-10, etc., and to reduce the rate of relapse. PE directly enhances muscle strength and cardiorespiratory fitness, as well as walking speed, endurance, and balance in MS patients. Furthermore, reductions in fatigue, symptoms of depression, and improvements in cognitive dysfunction and quality of life have been associated with PE in MS patients.

Despite the clear benefits of PE for MS patients, a significant proportion drop out or fail to maintain an active lifestyle post-rehabilitation. This tendency is a serious challenge for integrating and sustaining PE in the daily lives of individuals with MS. Consequently, the effectiveness of electronic health devices, or digital healthcare tools, in addressing the challenge remains an important area of interest. The effectiveness of new technology in MS rehabilitation, including telerehabilitation, has shown promising results in improving fitness, gait, balance, and upper limb function, often equaling or exceeding traditional methods.

It may be concluded that PE represents an effective therapeutic strategy for pwMS, however, further research is required to investigate PE's long-term impact on managing pwMS with comorbidities.

Study design This protocol delineates a prospective, longitudinal randomized controlled trial (RCT) aimed at evaluating the effects of an e-based PE intervention at home in addition to usual care on the disability progression of pwMS, both as an independent factor and in the context of comorbid conditions. Furthermore, an aim is to assess associations between PE and levels of inflammatory, metabolic, and neurodegenerative mediators and as well as clinical status, in pwMS with or without comorbidities.

Participants The study will include pwMS with T2DM as a well-defined and frequently occurring comorbidity, and pwMS without comorbidity. In addition, screening for vascular comorbidity and related risk factors as T2DM, hypertension and hyperlipidemia will be performed. The pwMS will be matched for age and gender as well as severity of disability. Details about the initiation and cessation of disease-modifying therapies (DMT) will be collected.

Blinding and Randomization procedure Patients will be randomized in a 1:1 ratio into groups receiving either usual care or usual care plus a 6-month e-Based PE program, using blocks of 4 or 6 by computer-generated assignment process. Patients in both groups will receive care as usual, which consist of single group therapy supervised by a physiotherapist 1 time a week. The extent of care the patient receives during the trial period will be registered. Due to the nature of the intervention, it is not feasible to blind participants or physiotherapists delivering the program. Nonetheless, to preserve the integrity of the trial, outcome assessors (researchers) will remain blinded to the allocation of treatments throughout the study.

Interventions The e-based exercise intervention comprises a 6-months home-based resistance training for the lower extremities, conducted twice weekly. The focus on the lower extremities is due to the marked impairment in muscle strength compared to the upper extremities in pwMS. The intervention adapts the principles of two previous studies on supervised machine-based resistance training for MS patients, which effectively improved walking performance. The original protocol is modified e-delivery, incorporating five exercises leg press, knee extension, hip flexion, hamstring curl, and hip extension-using resistance bands. While resistance band training has been beneficial for the upper extremity in MS in home-based training programs, its application to the lower extremity is to the best of our knowledge yet unproven.

All 48 sessions will be conducted in virtual groups of 6-8 participants, supervised by an experienced physiotherapist, connected to the virtual group from an exercise facility at the hospital using a 65" wide screen with computer hardware. The sessions will be hosted using Hospital-to-Citizen videoconference software.

Participants will perform exercises with a fast concentric phase and a slow eccentric phase.

Participants will initially receive both verbal and written instructions on using the online platform and have a one-on-one virtual session with the physiotherapist to test the setup. Resistance bands will be provided post-randomization. The sessions will be tested and proven feasible in a mixed-methods study in patients with chronic conditions. Additionally, a trial run will be conducted with a few patients with MS to optimize the procedure before the trial.

The self-management and exercise therapy program's details, including activities, duration, frequency, and methodologies, are documented following the Template for Intervention Description and Replication (TIDieR) and the Consensus on Exercise Reporting Template (CERT).

Comorbid conditions At the study outset comorbidity data, including diagnosis dates, characteristics, and treatments, will be extracted from patients' medical records, and supplemented by patient interviews as needed.

Cognitive assessment Participants' education level and hand preference will be assessed through interviews, and cognitive functions will be evaluated using the Montreal Cognitive Assessment (MoCA). Quality of life will be measured using the European Quality of Life-5 Dimensions (EQ-5D) index and visual analog scale (VAS), a range of scores from 0-100. A higher score indicates greater pain intensity.

Specimens Blood and cerebrospinal fluid (CSF) samples will be systematically collected at three key time points: baseline (prior to starting the exercise program), 6 months (upon completion of the program), at 12 and 24 months. All clinical and laboratory data derived from these samples will be analyzed while maintaining blinding to ensure unbiased assessment. The markers of inflammation, metabolism and neurodegeneration will be measured with sensitive assays.

MRI Participants will undergo initial and final CNS MRI using a 3 Tesla system will include brain, spinal cord, and optic nerve imaging with sequences like 3D FLAIR, T2 SPACE, and T1 MPRAGE. Advanced techniques like multi-parametric mapping and diffusion-weighted imaging will be employed for detailed CNS characterization, focusing on changes related to MS and vascular comorbidities.

Patient reported outcomes For assessing fatigue, the short-form Neuro-QOL Fatigue Scale will be utilized to measure current levels of fatigue. This scale provides a valuable insight into the impact of fatigue on the quality of life of participants. Health-related quality of life, assessed using the standardized 5-level EuroQol 5-dimensional questionnaire (EQ-5D-5L). Depression level was measured using the Personal Health Questionnaire Depression Scale (PHQ-8).

Outcome measures and assessment timeline Outcome measures will include the above-mentioned assessments, scheduled for documentation at baseline, 6, 12, and 24 months.

* Walking capacity, assessed by the Six-Minute Walk Test (6MWT) (unit: meter, higher numbers indicate better performance).
* Objective measurement of physical activity (PA) at baseline and study conclusion providing detailed data on PA patterns and intensities. Two accelerometers (m/s2) will be used to measure PA in each participant, who will wear two accelerometers attached to the skin with tape, one on the front of their thigh and one on the non-dominant wrist. Data will be analyzed by descriptions of daily- and weekly PA patterns and time spent on different activities with different intensity among participants before and after the intervention.
* Cognitive function, evaluated using the Montreal Cognitive Assessment (MoCA), a 30-item cognitive screen (higher numbers indicate better performance).
* Fatigue levels, assessed using the short-form Neuro-QOL Fatigue Scale (Units on a Scale, expressed as T scores with a mean of 50 and SD of 10).
* Disability progression, monitored by changes in the EDSS score (a scoring system between 0 and 10, the greater the level, the more disability) from baseline
* MRI new T2 lesion/enhancing lesion
* Number of MS Relapse(s)
* Adverse events (as detailed in section below)
* Body Mass Index (BMI) (weight /height, kg/meter2), blood pressure (mmHg), lipid profiles (triglyceride (mmol/l), HDL(mmol/l, HDL(mmol/l), , LDL(mmol/l), cholesterol(mmol/l),), fasting blood glucose (mmol/l), and insulin levels (mIU/L), glucose tolerance (mmol/l), and insulin resistance (Patients who require >1 unit/kg/day are considered to have insulin resistance).

Primary outcomes: We will evaluate walking capacity by 6MWT and the "no evidence of disease activity" (NEDA-3) score, which is characterized by three parameters, lack of clinical relapses and disease progression measured by EDSS and absence of new disease activity on MRI (new T2 lesions/enhancing lesion) over a period of observation time.

Secondary outcomes: Secondary outcomes include quality-of-life (MoCA) and fatigue (the short-form Neuro-QOL Fatigue Scale). Neurofilament Light Chain (NfL) levels will be used as marker of neuronal injury, unit pg/ml.

Adverse events Adverse events (AE) will be systematically documented for both the intervention and the usual care group using a patient diary over the course of the 6-month period. Patients will report any symptoms or pain experienced post-PE. Both AE and serious adverse events (SAE) will be proactively registered at all follow-up's visits, employing open-probe questioning to ensure comprehensive recording of all AEs. Additionally, patient medical records will be reviewed at the primary endpoint (6 months) to identify any AEs that have occurred since enrollment. AEs will be classified in accordance with the Food and Drug Administration's definition of an SAE. The recording, categorization, and assessment of the severity of AEs will be conducted irrespective of presumed causality with study treatments. These evaluations will be conducted at 3-, 6-, and 12-months post-intervention.

Data management The data related to this study will be securely stored in the REDCap database system. This approved electronic platforms is chosen for data collection and data storage to ensure that missing data are kept to a minimum and that privacy and confidentiality of personal data are maintained.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed MS diagnosis as per the 2017 MS criteria. [3]
2. Expanded Disability Status Scale (EDSS) assessment score of less than 7.0 at baseline.
3. Adults aged 18 years or above.
4. Commitment and mental ability to participate in a 6-month e-based physical exercise program, supervised bi-weekly by a physiotherapist.

Exclusion Criteria:

5. Change in prophylactic DMT within the last 3 months 6. Steroid treatment in the past month. 7. Drug or alcohol abuse. 8. Pregnancy. 9. Active systemic infection

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
6-meters' walk test | baseline, 6, 12, and 24 months
  Walking capacity, assessed by the 6-meters' walk test
"no evidence of disease activity" (NEDA-3) score | over a two years period of observation time
  The "no evidence of disease activity" (NEDA-3) score, which is characterized by three parameters, lack of clinical relapses and disease progression measured by EDSS and absence of new disease activity on MRI (new T2 lesions/enhancing lesion)

SECONDARY OUTCOMES:
Cognitive function, evaluated using the Montreal Cognitive Assessment (MoCA), | baseline, 6, 12, and 24 months
  cognitive function assessment (a 30-item cognitive screen (higher numbers indicate better performance).
Fatigue levels, assessed using the short-form Neuro-QOL Fatigue Scale | baseline, 6, 12, and 24 months
  Fatigue levels assessment (Units on a Scale, expressed as T scores with a mean of 50 and SD of 10).
Neurofilament Light Chain (NfL) determination | baseline, 6, 12, and 24 months
  NfL will be measured as marker of neuronal injury, unit pg/ml

CONTACTS AND LOCATIONS:
Overall Officials: Nasrin Asgari, Professor, Principal Investigator — Institute of Regional Health Research, University of Southern Denmark
Locations (1):
- University of Southern Denmark, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No